CLINICAL TRIAL: NCT02691910
Title: Efficacy of Chloroquine (CQ) Alone Compared to Concomitant CQ and Primaquine (PQ) for the Treatment of Uncomplicated Plasmodium Vivax Infection
Brief Title: Efficacy of Chloroquine (CQ) Alone Compared to Concomitant CQ and Primaquine for Plasmodium Vivax Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 404067/2012-3; 550.565 (Other: Ethics Committee of the Institute of Biomedical Sciences)
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Malaria, Vivax
Keywords: malaria; Plasmodium vivax; treatment; Chloroquine; Primaquine
MeSH Terms: conditions — Malaria, Vivax; Malaria | interventions — Chloroquine; chloroquine diphosphate; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONCURRENT CHLOROQUINE+PRIMAQUINE (Active Comparator): The infected individuals were treated with the standard chloroquine (CQ)+primaquine(PQ) regimen to malaria caused by Plasmodium vivax.
  * Chloroquine (tablet containing 150mg of base) - it was given on days 0 (10mg/kg), 1 (7.5mg/kg) and 2 (7.5mg/kg). Total dose, 25 mg base/kg.
  * Primaquine - it was given once a day (0.5 mg/kg) for seven days, starting on day 0 of CQ treatment. Total dose, 3.5mg/kg The medications were administered under direct observation and the patient was monitored for vomiting for 60 minutes.
  Interventions: Drug: Chloroquine; Drug: Primaquine
- CHLOROQUINE (Experimental): The infected individuals were initially treated with chloroquine (CQ) alone and the primaquine(PQ) was introduced on day 28.
  * Chloroquine (tablet containing 150mg of base) - it was given on days 0 (10mg/kg), 1 (7.5mg/kg) and 2 (7.5mg/kg). Total dose, 25 mg base/kg.
  * Primaquine - it was given once a day (0.5 mg/kg) for seven days, starting on day 28 of CQ treatment. Total dose, 3.5mg/kg.
  The medications were administered under direct observation and the patient was monitored for vomiting for 60 minutes.
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Chloroquine — 10mg/kg on day 0 and 7.5mg/kg on days 1 and 2. Total dose, 25 mg base/kg. Tablet containing 150mg of base.
  Other Names: Chloroquine diphosphate
Drug: Primaquine — 0.5 mg/kg once a day, for seven days. Total dose, 3.5mg/kg.
  Arms: CONCURRENT CHLOROQUINE+PRIMAQUINE

SUMMARY:
This is a randomized open-label trial to evaluate the efficacy of chloroquine (CQ) alone compared to chloroquine+primaquine (CQ+PQ) in the treatment of uncomplicated malaria caused by Plasmodium vivax infection in a endemic area in the westernmost part of the Amazon Basin of Brazil. The duration of follow up for evaluating CQ efficacy as a schizonticidal drug was 28 days. The duration of complete follow up to detect recurrent P. vivax infections by passive surveillance was six months. All patients in the CQ alone arm received 7 days of PQ treatment (3.5mg/kg total dose) starting on day 28 of the study follow-up.

DETAILED DESCRIPTION:
1. OBJECTIVE- To assess the efficacy of co-administered chloroquine+primaquine (CQ+PQ) vs.CQ alone (PQ being postponed up to day 28 of CQ therapy) as a schizontocidal therapy (28-day follow-up) and as radical cure among uncomplicated P. vivax malaria (6-month follow-up). Specifically:

   * To measure the clinical and parasitological efficacy of CQ+PQ vs. CQ alone, over 28 days of follow-up.
   * To measure the time to the first recurrent vivax malaria episode, between days 29 and 180 of follow-up.
2. METHODS - This is a randomized, open-label. The duration of follow up for evaluating CQ efficacy as a schizonticidal drug was 28 days. The duration of complete follow up to detect recurrent P. vivax infections by passive surveillance was six months. All patients in the CQ alone arm received 7 days of PQ (3.5mg/kg total dose) starting on day 28 of the follow-up.

   2.1 STUDY SITE AND POPULATION - The study was carried out in the city of Cruzeiro do Sul , Acre State, in the westernmost part of the Amazon Basin of Brazil. The study population was patients aged above 5 years diagnosed with uncomplicated P. vivax malaria, who gave permission for study inclusion.

   2.2 INCLUSION CRITERIA - mono-infection with P. vivax, age >5 years, ability to swallow oral medication, axillary temperature ≥37.5ºC (or history of fever in the last 48 hours) or to agree to comply with the study and provides written informed consent.

   2.3 EXCLUSION CRITERIA FOR ENROLLMENT - severe malaria requiring hospitalization, severe malnutrition (weight-for-age ≤ 3 standard deviations below the mean), co-infection with any other Plasmodium species, severe anemia (Hg<8g/100 ml), hypersensitivity to CQ or PQ, febrile conditions caused by diseases other than malaria, serious or chronic medical condition, pregnant or breastfeeding women, prior history of hemolysis or severe anemia or regular medication which may interfere with antimalarial pharmacokinetics.

   2.4 ENROLLMENT PROCEDURES 2.4.1. CLINICAL EVALUATION - All patients were evaluated for signs of febrile illness other than malaria, and signs of severe disease/danger in order to exclude the patient from participating in the study. Female of childbearing age was asked about pregnant and lactating. On screening and each subsequent visit, the patient was asked about fever in the last 48 hours and his/her current temperature was measured. Any disease/surgical conditions, drug allergies, use of medication or herbal supplements was recorded. The patient's pulse rate, respiratory rate, height, weight and the results of a baseline physical examination was recorded. This was done on screening and each subsequent visit.

   2.5. LABORATORY EVALUATIONS ON-SITE a - Urine β-HCG pregnancy test was conducted on women aged 13-49 b - Two thick blood smears were prepared on day 0 and at each follow-up visit (days 1, 2, 3, 7, 14, 21, 28, 180). One thick smears was examined on site to verify parasite species and a formal parasite count. The second slide was archived for later examination. Two qualified microscopists read all the slides independently. Discordant results were re-examined by a third microscopist, and parasite density was calculated by averaging the two closest counts. Microscopic diagnosis of malaria (parasite-specific DNA and gametocyte-specific RNA transcripts) was further confirmed by real-time quantitative PCR on days 0, 1, 2, 3, 28 and on the day of any parasite recurrence.

   c - Venous blood samples was collected on days 0, 1, 2, 3, 7, 28 and on the day of any parasite recurrence. It was used for on-site G6PD testing and a full blood count and hemoglobin measurement in addition to preparing thick smears. Plasma samples were stored at -80°C (or liquid nitrogen) and shipped to the central laboratory in São Paulo for immunological measurements (antibodies, cytokines). The remaining whole-blood aliquots were cryopreserved for DNA and RNA extraction and CQ measurements (the later on days 0 and 28 and on the day of any parasite recurrence). The whole-blood samples collected on day 0 and on the day of any parasite recurrence were cryopreserved for ex-vivo drug resistance assays.

   d - Finger-prick blood samples collected on days 14, 21, and 180 were used for hemoglobin measurements and to prepare thick smears. Remaining finger-prick blood samples were spotted onto FTA membranes for long-term DNA storage at 4°C.

   e - G6PD testing was conducted on-site on day 0. If the patient was G6PD deficient, she/he was excluded.

   2.6 SUBSEQUENT FOLLOW UP Each patient was clinically reassessed on days 1, 2, 3, 7, 14, 21, 28 and 180. Venous blood (days 1, 2, 3, 7, 28) or capillary (finger prick) blood samples (days 14, 21, 180) was examined for malaria parasites at each visit and on any other day if the patient spontaneously returns with fever or worsening symptoms.

   Hemoglobin status - measured on days 0, 1, 2, 3, 7, 14, 21, 28, 180, and on the day of any parasite recurrence.

   Drug level testing- venous blood should be collected on days 0, 7, 28 and on the day of recurrent parasitemia to measure concentrations of CQ.

   Molecular testing - P. vivax isolates from recurrent infections up to day 28 would be genotypically compared with those from day 0 using a panel of 14 highly polymorphic microsatellite markers in order to determine whether the recurrence is due to the only or major parasite population present in the original infection, to a minor parasite subpopulation that could be detected on day 0 or to a completely different parasite population.

   2.7 TREATMENT All participants received CQ (total dose, 25 mg base/kg) and PQ (total dose, 3.5mg/kg) supervised by a study nurse.

   CQ: on days 0 (10mg/kg), 1 and 2 (7.5mg/kg). PQ: once a day (0.5 mg/kg) for seven days, starting either on day 0 of CQ treatment (concurrent CQ-PQ treatment arm) or on day 28 (CQ alone arm).

   2.8 FOLLOW-UP PROCEDURES 2.8.1. Active Surveillance - Study participants were visited on days 0, 1, 2, 3, 7, 14, 21, 28, and 180. At each visit, a questionnaire was completed asking about history or fever currently or in the preceding month and a venous or capillary sample was collected for blood slide examination and to check for parasitemia.

   2.8.2. Passive Surveillance - Patients were advised to return to the health center on any day if symptoms, sign of danger (unable to drink or breastfeed, vomiting everything, presenting with convulsions, lethargic or unconscious, unable to sit or stand, presenting with difficult breathing), if they are still sick or if there is any cause for worry. During the period of PQ administration, anyone reporting dark urine or abdominal cramps (signs of toxicity) should seek medical attention.

   2.8.3. Rescue treatment - A recurrent vivax parasitaemia within 28 days is potentially a recrudescent infection. These patients would be re-treated with the standard CQ-PQ co-administration regimen and remain in the study. After 28 days, a recurrent vivax parasitaemia is more likely a relapse or a new infection. These patients would be treated with the standard CQ-PQ co-administration regimen. Patients who develop severe malaria would be admitted to hospital and treated according to the guidelines of the Ministry of Health of Brazil.

   2.8.4. Discontinuation/Withdrawal of Participants from Study Treatment Each participant had the right to withdraw from the study at any time. The investigator would withdraw a participant if the participant had blood transfusion or a fall in Hb to less than 7g/dL or a macroscopic haemoglobinuria or a fall in Hb by >25% (within the first 14 days or 8 weeks, as above) or significant protocol deviation, disease progression, lost of follow up, use of drugs with antimalarial activity, an important adverse event or an emergency event.
3. END-POINTS 3.1 Schizontocidal Efficacy of Chloroquine It was derived by the risk of recurrence until day 28 in the CQ only arm.

   * Schizontocidal Therapeutic Failure (TF): clinical deterioration which requires hospitalization in the presence of asexual parasitemia OR asexual parasitemia with temperature > 37.5°C between days 3 and 28 OR parasitemia between days 7 and 28, irrespective of the clinical condition.
   * Adequate Schizontocidal Response (ACR): absence of parasitemia on days 7, 14, 21 and 28 without previously meeting the criteria of TF.

   3.2 Safety end points The main concern with PQ lies in the risk of severe hemolytic reactions, and a fall in haemoglobin. However, decreasing hemoglobin can also occur following P. vivax malaria. It is therefore vital to monitor for evidence of hemolysis and clinical significant fall in Hb. Hemoglobin concentration was assessed on days 0, 1, 2, 3, 7, 14, 21, 28, and 180, with the lowest levels expected from day 3 to 14.

   3.2.1.Adverse Event (AE): Any unfavourable and unintended sign, symptom or disease temporally associated with the use of the study medication, without necessarily a causal relationship.

   3.2.2.Adverse Reaction (AR). An untoward and unintended sign, symptom or disease judged as having a suspected causal relationship to the study medication.

   3.2.3.Serious Adverse Event (SAE). Any untoward medical occurrence that at any dose results in death or risk of death, requires hospitalization, results in persistent or significant disability/incapacity.
4. STATISTICAL ANALYSIS The primary outcome and the safety data were analyzed on a modified intention-to-treat population. A conservative analysis will be repeated on the per protocol population excluding patients with subsequent major protocol violations. The primary outcome will be the proportion of therapeutic failure observed up to day 28 of follow-up in each study arm. The investigators will compare the cumulative incidence of P. vivax recurrence between study arms. SPSS version 17.0 will be used for data management and analysis. Data will be analyzed by Kaplan-Meier (KM) method and per-protocol analysis. The time to the first parasite recurrence within 28 days of follow-up (primary outcome) and between days 29 and 180 (secondary outcome) will be calculated using KM estimates (survival analysis). Statistical comparisons will be made between the arms using the log rank test. The proportions of clinical and parasitological failure, and adequate clinical and parasitological response at day 28 will be calculated, with their respective 95% confidence intervals.
5. ETHICAL ISSUES - The study were fully explained to the participants and ask for their consent/assent to participate. Consenting participants might terminate their participation at any time. All case record forms were accessed only by authorized staff members. Participants were informed of the results of the exams and clinical assessments at each follow-up visit.
6. DEFINITION OF TREATMENT OUTCOMES

   * Early treatment failure (ETF)

     * danger signs or severe malaria on day 1, 2 or 3 in the presence of parasitaemia
     * parasitaemia on day 2 higher than on day 0, irrespective of axillary temperature
     * parasitaemia on day 3 with axillary temperature ≥ 37.5 ºC
     * parasitaemia on day 3 ≥25% of count on day 0
   * Late treatment failure
   * Late clinical failure (LCF)

     * danger signs or severe malaria in the presence of parasitaemia on any day between day 4 and day 28 in patients who did not previously meet any of the criteria of early treatment failure
     * parasitaemia on any day between day 4 and day 28 with axillary temperature ≥37.5ºC (or history of fever) in patients who did not previously meet any of the criteria of early treatment failure
   * Late parasitological failure (LPF) - Parasitaemia on any day between day 7 and day 28 with axillary temperature <37.5ºC in patients who did not previously meet any of the criteria of early treatment failure or late clinical failure.
   * Adequate clinical and parasitological response - Absence of parasitaemia on day 28, irrespective of temperature, in patients who did not previously meet any of the criteria of ETF, LCF or LPF.

ELIGIBILITY:
Inclusion Criteria:

* Slide-confirmed mono-infection with P. vivax
* Age > 5 years
* Ability to swallow oral medication
* Axillary temperature ≥ 37.5º C or history of fever during the previous 48 hours
* Patient or caregiver agrees to comply with the study protocol (including blood collections and return visits) and provides written informed consent.

Exclusion Criteria:

* General danger signs or symptoms of severe malaria requiring hospitalization
* Signs or symptoms of severe malnutrition, defined as weight-for-age ≤ 3 standard deviations below the mean (NCHS/WHO normalized reference values)
* Slide-confirmed co-infection with any other Plasmodium species
* Severe anemia, defined as Hg<8g/100 ml
* Known hypersensitivity to any of the drugs being evaluated
* Presence of febrile conditions caused by diseases other than malaria
* Serious or chronic medical condition by history (cardiac, renal, hepatic diseases, sickle cell disease, HIV/AIDS)
* Pregnant or breastfeeding women
* Prior history of hemolysis or severe anemia
* Regular medication which may interfere with antimalarial pharmacokinetics

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Early treatment failure | within the first 3 days
  danger signs or severe malaria on day 1, 2 or 3 in the presence of parasitaemia OR parasitaemia on day 2 higher than on day 0 OR parasitaemia on day 3 with axillary temperature ≥ 37.5 ºC OR parasitaemia on day 3 ≥ 25% of count on day 0

SECONDARY OUTCOMES:
Late clinical failure | 28 days
  danger signs or severe malaria in the presence of parasitaemia on any day between day 4 and day 28 OR parasitaemia on any day between day 4 and day 28 with axillary temperature ≥ 37.5 ºC (or history of fever) in patients who did not previously meet any of the criteria of early treatment failure
Late parasitological failure | 28 days
  presence of parasitaemia on any day between day 7 and day 28 with axillary temperature < 37.5 ºC in patients who did not previously meet any of the criteria of early treatment failure or late clinical failure

OTHER OUTCOMES:
Adverse Event | 180 days
  Any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of the study medication, whether or not considered related to the study medication.
Adverse Reaction | 180 days
  Any untoward and unintended responses to a medicinal product related to any dose judged by either the reporting medically qualified professional or the sponsor as having a reasonable suspected causal relationship to the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: MARCELO U FERREIRA, MD-PHD, Study Director — Biomedical Sciences Institute of São Paulo University; SIMONE L ANDRADE, MD-PHD, Principal Investigator — Oswaldo Cruz Institute
Locations (2):
- Brazil (2):
  - Oswaldo Cruz Foundation, Rio de Janeiro, Rio de Janeiro
  - Institute of Biomedical Sciences, University of Sao Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez G, Pineros JG, Tobon A, Rios A, Maestre A, Blair S, Carmona-Fonseca J. Efficacy of three chloroquine-primaquine regimens for treatment of Plasmodium vivax malaria in Colombia. Am J Trop Med Hyg. 2006 Oct;75(4):605-9. PMID 17038680
- [Background] Anez A, Navarro-Costa D, Yucra O, Garnica C, Melgar V, Moscoso M, Arteaga R, Nakao G. [Therapeutic response of Plasmodium vivax to chloroquine in Bolivia]. Biomedica. 2012 Oct-Dec;32(4):527-35. doi: 10.1590/S0120-41572012000400008. Spanish. PMID 23715228
- [Background] Arias AE, Corredor A. Low response of Colombian strains of Plasmodium vivax to classical antimalarial therapy. Trop Med Parasitol. 1989 Mar;40(1):21-3. PMID 2662351
- [Background] Baird JK. Resistance to therapies for infection by Plasmodium vivax. Clin Microbiol Rev. 2009 Jul;22(3):508-34. doi: 10.1128/CMR.00008-09. PMID 19597012
- [Background] Baird JK, Leksana B, Masbar S, Fryauff DJ, Sutanihardja MA, Suradi, Wignall FS, Hoffman SL. Diagnosis of resistance to chloroquine by Plasmodium vivax: timing of recurrence and whole blood chloroquine levels. Am J Trop Med Hyg. 1997 Jun;56(6):621-6. doi: 10.4269/ajtmh.1997.56.621. PMID 9230792
- [Background] Baird KJ, Maguire JD, Price RN. Diagnosis and treatment of Plasmodium vivax malaria. Adv Parasitol. 2012;80:203-70. doi: 10.1016/B978-0-12-397900-1.00004-9. PMID 23199489
- [Background] Baird JK, Tiwari T, Martin GJ, Tamminga CL, Prout TM, Tjaden J, Bravet PP, Rawlins S, Ferrel M, Carucci D, Hoffman SL. Chloroquine for the treatment of uncomplicated malaria in Guyana. Ann Trop Med Parasitol. 2002 Jun;96(4):339-48. doi: 10.1179/000349802125001023. PMID 12171615
- [Background] Bray PG, Deed S, Fox E, Kalkanidis M, Mungthin M, Deady LW, Tilley L. Primaquine synergises the activity of chloroquine against chloroquine-resistant P. falciparum. Biochem Pharmacol. 2005 Oct 15;70(8):1158-66. doi: 10.1016/j.bcp.2005.07.021. PMID 16139253
- [Background] Carmona-Fonseca J, Maestre A. Prevention of Plasmodium vivax malaria recurrence: efficacy of the standard total dose of primaquine administered over 3 days. Acta Trop. 2009 Nov;112(2):188-92. doi: 10.1016/j.actatropica.2009.07.024. Epub 2009 Aug 3. PMID 19653988
- [Background] Castillo CM, Osorio LE, Palma GI. Assessment of therapeutic response of Plasmodium vivax and Plasmodium falciparum to chloroquine in a Malaria transmission free area in Colombia. Mem Inst Oswaldo Cruz. 2002 Jun;97(4):559-62. doi: 10.1590/s0074-02762002000400020. PMID 12118291
- [Background] de Santana Filho FS, Arcanjo AR, Chehuan YM, Costa MR, Martinez-Espinosa FE, Vieira JL, Barbosa Md, Alecrim WD, Alecrim Md. Chloroquine-resistant Plasmodium vivax, Brazilian Amazon. Emerg Infect Dis. 2007 Jul;13(7):1125-6. doi: 10.3201/eid1307.061386. No abstract available. PMID 18214203
- [Background] Egan TJ. Chloroquine and primaquine: combining old drugs as a new weapon against falciparum malaria? Trends Parasitol. 2006 Jun;22(6):235-7. doi: 10.1016/j.pt.2006.03.006. Epub 2006 Apr 3. PMID 16580880
- [Background] Garavelli PL, Corti E. Chloroquine resistance in Plasmodium vivax: the first case in Brazil. Trans R Soc Trop Med Hyg. 1992 Mar-Apr;86(2):128. doi: 10.1016/0035-9203(92)90535-k. No abstract available. PMID 1440766
- [Background] Marques MM, Costa MR, Santana Filho FS, Vieira JL, Nascimento MT, Brasil LW, Nogueira F, Silveira H, Reyes-Lecca RC, Monteiro WM, Lacerda MV, Alecrim MG. Plasmodium vivax chloroquine resistance and anemia in the western Brazilian Amazon. Antimicrob Agents Chemother. 2014;58(1):342-7. doi: 10.1128/AAC.02279-12. Epub 2013 Oct 28. PMID 24165179
- [Background] Naing C, Aung K, Win DK, Wah MJ. Efficacy and safety of chloroquine for treatment in patients with uncomplicated Plasmodium vivax infections in endemic countries. Trans R Soc Trop Med Hyg. 2010 Nov;104(11):695-705. doi: 10.1016/j.trstmh.2010.08.009. Epub 2010 Sep 20. PMID 20850161
- [Background] Osorio L, Perez Ldel P, Gonzalez IJ. [Assessment of the efficacy of antimalarial drugs in Tarapaca, in the Colombian Amazon basin]. Biomedica. 2007 Mar;27(1):133-40. Epub 2007 May 31. Spanish. PMID 17546230
- [Background] Phillips EJ, Keystone JS, Kain KC. Failure of combined chloroquine and high-dose primaquine therapy for Plasmodium vivax malaria acquired in Guyana, South America. Clin Infect Dis. 1996 Nov;23(5):1171-3. doi: 10.1093/clinids/23.5.1171. PMID 8922821
- [Background] Rieckmann KH, Davis DR, Hutton DC. Plasmodium vivax resistance to chloroquine? Lancet. 1989 Nov 18;2(8673):1183-4. doi: 10.1016/s0140-6736(89)91792-3. PMID 2572903
- [Background] Ruebush TK 2nd, Zegarra J, Cairo J, Andersen EM, Green M, Pillai DR, Marquino W, Huilca M, Arevalo E, Garcia C, Solary L, Kain KC. Chloroquine-resistant Plasmodium vivax malaria in Peru. Am J Trop Med Hyg. 2003 Nov;69(5):548-52. PMID 14695094
- [Background] Russell B, Chalfein F, Prasetyorini B, Kenangalem E, Piera K, Suwanarusk R, Brockman A, Prayoga P, Sugiarto P, Cheng Q, Tjitra E, Anstey NM, Price RN. Determinants of in vitro drug susceptibility testing of Plasmodium vivax. Antimicrob Agents Chemother. 2008 Mar;52(3):1040-5. doi: 10.1128/AAC.01334-07. Epub 2008 Jan 7. PMID 18180357
- [Background] Russell BM, Udomsangpetch R, Rieckmann KH, Kotecka BM, Coleman RE, Sattabongkot J. Simple in vitro assay for determining the sensitivity of Plasmodium vivax isolates from fresh human blood to antimalarials in areas where P. vivax is endemic. Antimicrob Agents Chemother. 2003 Jan;47(1):170-3. doi: 10.1128/AAC.47.1.170-173.2003. PMID 12499187
- [Background] Soto J, Toledo J, Gutierrez P, Luzz M, Llinas N, Cedeno N, Dunne M, Berman J. Plasmodium vivax clinically resistant to chloroquine in Colombia. Am J Trop Med Hyg. 2001 Aug;65(2):90-3. doi: 10.4269/ajtmh.2001.65.90. PMID 11508397
- [Background] Villalobos-Salcedo JM, Tada MS, Kimura E, Menezes MJ, Pereira da Silva LH. In-vivo sensitivity of Plasmodium vivax isolates from Rond nia (western Amazon region, Brazil) to regimens including chloroquine and primaquine. Ann Trop Med Parasitol. 2000 Dec;94(8):749-58. doi: 10.1080/00034980020027960. PMID 11214093
- [Derived] Ladeia-Andrade S, Menezes MJ, de Sousa TN, Silvino ACR, de Carvalho JF Jr, Salla LC, Nery OA, de Melo GNP, Corder RM, Rodrigues PT, Ferreira MU. Monitoring the Efficacy of Chloroquine-Primaquine Therapy for Uncomplicated Plasmodium vivax Malaria in the Main Transmission Hot Spot of Brazil. Antimicrob Agents Chemother. 2019 Apr 25;63(5):e01965-18. doi: 10.1128/AAC.01965-18. Print 2019 May. PMID 30782991